CLINICAL TRIAL: NCT06564025
Title: Pilot of a Father-based Intervention to Support Adolescents' Reproductive Health
Brief Title: Pilot of an Online Sexual Health Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wellesley College (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jennifer Grossman, Principal Investigator, Wellesley College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23139; 1R21HD109744-01A1 (NIH)
Record Dates: First submitted 2024-08-02; First posted 2024-08-21 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Program, Communication
Keywords: sex education; father-teen program; family intervention
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: To assess program feasibility, acceptability, and preliminary efficacy, the investigators will pilot the intervention with a purposive sample of 50 father-teen pairs. All participants will receive the intervention. An online screener, pre- and post-intervention surveys, and brief module feedback will assess feasibility and acceptability. Pre- and post-intervention surveys will provide initial data on directionality for correlates of teens' sexual risk behaviors to determine whether a full-scale R01 is warranted. Debrief interviews with a purposive sample of pilot participants (5 fathers, 5 teens) will obtain in-depth intervention feedback and conduct member checks on module feedback. The investigators will revise the intervention prototype based on feasibility, acceptability, and preliminary efficacy data, then write up and distribute findings for dissemination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot group for program (Experimental): To assess program feasibility, acceptability, and preliminary efficacy, we will pilot the intervention with a purposive sample of 50 father-teen pairs (100 participants total). All participants will receive the program.
  Interventions: Behavioral: Pilot program study

INTERVENTIONS:
Behavioral: Pilot program study — To assess program feasibility, acceptability, and preliminary efficacy, we will pilot the intervention with a purposive sample of 50 father-teen pairs (100 participants total). All participants will receive the program.

SUMMARY:
This study proposes to pilot an online intervention to support father-teen health-promoting talk about sex and relationships using Social Cognitive Theory, and to evaluate this intervention's acceptability, feasibility, and preliminary efficacy, using an Intervention Mapping approach. This study involves conducting a pilot intervention with 50 pairs of fathers and their high-school aged teens. Feasibility and acceptability will be assessed through program data such as participants' pilot enrollment, lesson feedback, and program retention, survey data and member checks through debrief interviews (5 father, 5 teens). Preliminary assessment of directionality of change in participants' health-related knowledge, self-efficacy, and outcome expectations over the course of the pilot intervention (pre- and post-intervention surveys) to determine whether a full-scale R01 is warranted.

DETAILED DESCRIPTION:
This study proposes to pilot an online intervention to support father-teen health-promoting talk about sex and relationships using Social Cognitive Theory, and to evaluate this intervention's acceptability, feasibility, and preliminary efficacy, using an Intervention Mapping approach. This study involves conducting a pilot intervention with 50 pairs of fathers and their high-school aged teens. Feasibility and acceptability will be assessed through program data such as participants' pilot enrollment, lesson feedback, and program retention, survey data from Acceptability of Intervention Measure and Feasibility of Intervention Measure, and member checks through debrief interviews (5 father, 5 teens). Preliminary assessment of directionality of change in participants' health-related knowledge, self-efficacy, and outcome expectations over the course of the pilot intervention (pre- and post-intervention surveys) to determine whether a full-scale R01 is warranted.

The investigators will recruit a diverse sample of father-adolescent pairs (N=50 pairs) through partnership with three community partner organizations. Fathers will be asked questions online to determine project eligibility and demographics (screener) and given an online consent form. If a father agrees to teens' participation, the teen will be sent an assent form for their own participation and a brief screener survey. If teens are 18 or older, the investigators will request their contact information from participating fathers and ask teens to provide their own consent. Only father/teen pairs who complete the screeners and consent/assent forms, meet eligibility criteria, and both agree to participate can join the study.

All pilot participants will be given a pre-and post-intervention survey to assess any change in proximal outcomes. Participants will be asked to participate in 3 online modules over 6 weeks which include 3 online lessons (father and teens complete separately) and father/teen activities (fathers and teens complete together) and 3 father support group (father only). Each module will last one week and will include an online lesson and father-teen activity (fathers and teens) and online father support group session (fathers only). Lessons and support group sessions will include feedback questions (acceptability). Tracking of enrollment, retention, and duration of lesson participation will provide feasibility assessment. To obtain in-depth feedback on participants' responses to the intervention (acceptability), and to conduct member checks on pilot lesson feedback, the investigators will conduct debrief interviews with a purposive sample of pilot participants (5 fathers, 5 teens) with variation in: teen gender and level of intervention engagement.

The 3 module, 3-week intervention will be delivered on Qualtrics and Zoom, accessible via computer or tablet. Online lessons will be self-paced within each week and will each include a father-teen activity, with text and e-mail reminders at the start and end of the week. Father support groups will occur online at a scheduled time planned based on fathers' schedules. Given the limited scope of the project, prototype technology will be relatively simple, with more advanced technology planned for a future R01.

ELIGIBILITY:
Inclusion criteria for fathers:

* adult (18 or older)
* father (biological, step, adopted, or foster) of a participating teen and
* report regular contact with the teen
* healthy enough to participate in online surveys, an online intervention, interactive activities (either online, over the phone or in-person) with the adolescent, and an online support group
* speak English
* have a reading level of 6th grade or above.

Exclusion criteria for fathers:

* not a father (biological, step, adopted, or foster) of a participating high-school aged teen
* under the age of 18
* not in regular contact with their teen
* cannot participate in intervention in English Inclusion criteria for adolescents
* high-school aged child (biological, step, adopted, or foster) of a participating father
* report regular contact with their father
* healthy enough to participate in online surveys and interactive activities (either online, over the phone or in-person) with the father
* have a reading level of 6th grade or above Exclusion criteria for adolescents
* not in high school
* not in regular contact with the father
* not child (biological, step, adopted, or foster) of participating father
* cannot participate in intervention in English

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sexual knowledge | immediately before and immediately after the intervention
  Participants' knowledge about contraception, condom use, and sexually transmitted infections for fathers and teens (3 sub-scales, self-report, true/false with higher score indicating greater knowledge).
Sexual Communication Self-Efficacy Scale | immediately before and immediately after the intervention
  Teen participants' confidence in their capacity to talk with a partner about sexual issues including using protection during sex (5 subscales, self-report, 4-point Likert scales with 1-4 score range with higher scores indicating higher self-efficacy).
Self-Efficacy in Relationships | immediately before and immediately after the intervention
  Teen participants' confidence in their capacity to talk with a partner what they want and do not want in a relationship such as breaking up with someone they no longer like (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating higher self-efficacy).
Self-Efficacy for Consent | immediately before and immediately after the intervention
  Teen participants' confidence in their capacity to talk with a partner about consent, including asking for consent for sex (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating higher self-efficacy).
Self-Efficacy for Communication with Teens about Sex | immediately before and immediately after the intervention
  Father participants' confidence in their capacity to talk with their teen about sexual issues and relationships (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating higher self-efficacy).
Comfort Talking with Family about Sex | immediately before and immediately after the intervention
  Participants' comfort to talk with their father/teen about sexual issues and relationships for fathers and teens including being able to talk openly and honestly about sex (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating higher comfort).
Open Communication Scale | immediately before and immediately after the intervention
  Participants' comfort to talk with their father/teen about sex and relationships for fathers and teens including comfort talking through questions about sex (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating higher comfort).
Communication about Sex and Protection | immediately before and immediately after the intervention
  Participants' reported frequency of talk with their father/teen about sex and relationships including talking with your father/teen about how to use condoms (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating more frequent communication).
Communication with family about sex & relationships | immediately before and immediately after the intervention
  Participants' reported frequency of talk with their father/teen about sex and relationships including talk about value about sex and relationships (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating more frequent communication).
Frequency of Talk with Family about Sex and Relationships | immediately before and immediately after the intervention
  Participants' reported frequency of talk with their father/teen about sex and relationships including when it is ok to have sex (self-report, 4-point Likert scales with 1-4 score range with higher scores indicating more frequent communication).
Feasibility of Intervention Measure | immediately after the intervention
  Participants' experience of the program's accessibility including whether the program seems doable for fathers and teens (self-report, 5-point Likert scales with 1-5 score range with higher scores indicating higher feasibility).
Feasibility: Participants' experience of the program's ease | immediately after the intervention
  Participants' experience of the program's ease of use including whether the program was well-organized for fathers and teens (self-report, 5-point Likert scales with 1-5 score range with higher scores indicating higher feasibility).
Acceptability of Intervention Measure: whether participants approve of the program | immediately after the intervention
  Participants' experience of the program including whether they approve of the program for fathers and teens (self-report, 5-point Likert scales with 1-5 score range with higher scores indicating higher acceptability).
Intervention Acceptability and Tolerability: Participants' experience of the program's importance | immediately after the intervention
  Participants' experience of the program's importance including whether they think the program was helpful for fathers and teens (self-report, 5-point Likert scales with 1-5 score range with higher scores indicating higher acceptability).

CONTACTS AND LOCATIONS:
Locations (1):
- Wellesley College, Wellesley, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Documentation to be made publicly available to the research community will include pilot surveys and interview protocols, along with a detailed User Guide for interviews. A survey codebook will include a description of all items and survey measures as well as variable names, variable labels, and standard codes for missing values. Interview data will include a description of recoded data categories. We expect study data and associated documentation will be made available to the research community free of charge through the Inter-university Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol
Time Frame: Final submission and release of the study data will occur approximately 1 year following the end of fieldwork. Study data deposited in the Inter-university Consortium for Political and Social Research will be available to the research community in perpetuity. Datasets underlying methodological publications will be shared at or prior to initial publication date as appropriate.
Access Criteria: Deidentified pilot survey data will be made available as public use data to the research community via the Inter-university Consortium for Political and Social Research (ICPSR). Users of this data must register with ICPSR and agree to the Terms of Use. Data users also agree not to share or redistribute any data downloads.
  Recoded interview data that is determined to be potentially identifying through indirect or deductive disclosure are provided under restricted data contract to users who demonstrate a valid research need and meet conditions of use.